CLINICAL TRIAL: NCT01299623
Title: Disseminating Breast Cancer Prevention to African American Women
Brief Title: Breast Cancer Prevention Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 1R18HSO19339-01
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer Prevention
Keywords: breast cancer; breast cancer prevention; African American women
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evidential Group (Active Comparator): Participants in this group will receive education about breast cancer prevention and specific information about African American women and breast cancer risk.
  Interventions: Behavioral: Comparison of evidential versus non-evidential education on women's breast cancer prevention behaviors
- Non-Evidential Group (Active Comparator): Participants in this group will receive general information about breast cancer prevention without anything specific to African American women.
  Interventions: Behavioral: Comparison of evidential versus non-evidential education on women's breast cancer prevention behaviors

INTERVENTIONS:
Behavioral: Comparison of evidential versus non-evidential education on women's breast cancer prevention behaviors — Participants will be randomized to either the evidential or non-evidential group. Both groups will receive primarily the same information, except one group will receive information that is more tailored to African American women, while participants in the other group will receive general information about breast cancer prevention.

SUMMARY:
We will develop and evaluate a community-based approach for disseminating comparative effective reviews (CERs) about breast cancer prevention to African American women. The specific aims of our research, as shown below, will target this population because of persistent disparities in breast cancer morbidity and mortality among this population. Our primary aims are:

1. To evaluate uptake of a community-based strategy for disseminating CERs about breast cancer prevention to African American women based on sociodemographic characteristics, beliefs about medical research, and medical history. We predict that participation in a community forum will be higher among women with greater socioeconomic resources, those who have a family history of breast cancer, and women who have more positive beliefs about research.
2. To evaluate the impact of evidential versus non-evidential content about breast cancer prevention on psychological and behavioral outcomes that include: knowledge of breast cancer risk factors and prevention strategies, communication with individuals in their social and medical network, and distrust of medical research. We predict that women who receive evidential content that is specific for African American women will report greater knowledge about breast cancer risk factors and prevention strategies, will be more likely to discuss breast cancer prevention strategies with individuals in their social and medical network, and will report greater reductions in distrust of medical research compared to those who receive non-evidential content.

ELIGIBILITY:
Inclusion Criteria:

* African American women
* Ages 35-70
* No personal history of cancer
* Resident of Philadelphia metropolitan area

Exclusion Criteria:

* Non-African American
* Male
* Under 35 or over 70 years of age
* Personal history of cancer
* Not a resident of Philadelphia Metropolitan Area

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2010-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Intervention uptake | 1 session
  Assessment of participants' attendance at a session.
knowledge about breast cancer prevention | 6 months
  Measurement of women's knowledge about breast cancer prevention at three and six months post intervention compared to baseline measurements.
Communication about breast cancer prevention | 6 months
  Assessment of the extent to which women discuss breast cancer prevention with their health care providers at three and six months post intervention compared to at baseline.
Distrust of medical research | 6 months
  Assessment of the extent to which participants harbor distrust for the medical establishment three and six months post intervention compared to at baseline.

SECONDARY OUTCOMES:
Education | baseline
  Assessment of the relationship between participants' education and primary outcomes.
Family history | baseline
  Assessment of the relationship between participants' family history and the primary outcomes.
Beliefs about research | baseline
  Assessment of the relationship between participants' beliefs about research and the primary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Chanita H Halbert, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Community Based Research and Health Disparities, Philadelphia, Pennsylvania, United States